CLINICAL TRIAL: NCT03357380
Title: A Trial Investigating the Effect of Subcutaneous Semaglutide on Liver Fibrosis Assessed by Magnetic Resonance Elastography in Subjects With Non-alcoholic Fatty Liver Disease
Brief Title: A Study on How Semaglutide Works on Early Stages of Scar Tissue in the Liver Assessed by Pictures of the Liver
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9931-4381; 2017-001193-42 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1194-3900 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Hepatobiliary Disorders; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Digestive System Diseases; Non-alcoholic Fatty Liver Disease | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide (Experimental): Semaglutide will be initiated with a starting dose of 0.05 mg/day for the first 4 weeks. The dose will be increased every 4 weeks until the target dose of 0.4 mg/day has been reached.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Placebo will be initiated with a starting volume corresponding to 0.05 mg/day of semaglutide for the first 4 weeks. The volume will then be increased every 4 weeks until the target volume corresponding to 0.4 mg/day of semaglutide has been reached.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Subcutaneously (under the skin) once-daily. Will be increased more or less every 4 weeks. It is expected that from week 16 until week 72 The participants take the maximum planned dose (0.4 mg) of study medicine.
  Arms: Semaglutide
Drug: Placebo — Subcutaneously (under the skin) once-daily. Will be increased more or less every 4 weeks. It is expected that from week 16 until week 72 The participants take the maximum planned dose (0.4 mg) of study medicine.
  Arms: Placebo

SUMMARY:
This study is looking at the effect of semaglutide on subjects with nonalcoholic fatty liver disease.This study is comparing the change in early stages of scar tissue in the liver and fat deposition in the liver in people taking semaglutide and placebo (a dummy medicine).

Participants will either get semaglutide or placebo; which treatment participants get is decided by chance. Semaglutide is a medicine under clinical investigation. That means that the medicine has not yet been approved by the authorities. Participants will need to self-inject medicine once daily for 72 weeks. The medicine should be injected under the skin in the stomach, thigh or upper arm.

There are about 3 weeks before participants start the study medicine and 7 weeks after you stop it. The study will last for about 82 weeks in total.

Participants will have 12 clinic visits, 6 phone calls and 4 visits to an MRI centre.

The study includes MRI scans of the stomach. The MRI scans will take place at a different location. Participants will be excluded from the study if the study doctor thinks that there are risks for participants health. Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, aged 18-75 years (both inclusive) at the time of signing informed consent
* Liver steatosis greater than or equal to 10% measured by magnetic resonance imaging proton density fat fraction at screening
* Liver stiffness between 2.50 and 4.63 kPa (both inclusive) measured by magnetic resonance elastography at screening
* Body mass index between 25.0 and 40.0 kg/sqm (both inclusive) at the screening visit

Exclusion Criteria:

* Known or suspected abuse of alcohol (greater than 12 g/day for women or greater than 24 g/day for men) or alcohol dependence assessed by the Alcohol Use Disorders Identification Test (AUDIT questionnaire)
* Diagnosis of type 1 diabetes according to medical records
* Glycosylated haemoglobin A1c (HbA1c) greater than 9.5% at screening
* History or presence of pancreatitis (acute or chronic) as declared by the subject
* Screening calcitonin greater than or equal to 100 ng/L
* Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma (as declared by the subject)
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using highly effective contraceptive methods. (Highly effective contraceptive methods are considered those with a failure rate less than 1% undesired pregnancies per year including surgical sterilisation, hormonal intrauterine devices (coil), oral hormonal contraceptives, sexual abstinence (only acceptable if corresponding to the preferred and usual lifestyle of the subject) or a surgically sterilised partner)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Change in liver stiffness (kPa) assessed by magnetic resonance elastography (MRE) | Up to day -20, week 48
  Measured in KPa

SECONDARY OUTCOMES:
Change in liver stiffness (kPa) assessed by magnetic resonance elastography (MRE) | Up to day -20, week 24
  Measured in KPa
Change in liver stiffness (kPa) assessed by magnetic resonance elastography (MRE) | Up to day -20, week 72
  Measured in KPa
Change in relative liver fat content (%) assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | Up to day -20, week 24
  Measured in Percentage (%)
Change in relative liver fat content (%) assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | Up to day -20, week 48
  Measured in Percentage (%)
Change in relative liver fat content (%) assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | Up to day -20, week 72
  Measured in Percentage (%)
Change in absolute liver fat volume (L) assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | Up to day -20, week 24
  Measured in Percentage (%)
Change in absolute liver fat volume (L) assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | Up to day -20, week 48
  Measured in L
Change in absolute liver fat volume (L) assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | Up to day -20, week 72
  Measured in L
Proportion of subjects with at least 30% reduction in relative liver fat content assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | Weeks 0 - 24
  Number of subjects
Proportion of subjects with at least 30% reduction in relative liver fat content assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | Weeks 0 - 48
  Number of subjects
Proportion of subjects with at least 30% reduction in relative liver fat content assessed by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | Weeks 0 - 72
  Number of subjects
Proportion of subjects with at least 15% reduction in liver stiffness assessed by magnetic resonance elastography (MRE) | Weeks 0 - 24
  Number of subjects
Proportion of subjects with at least 15% reduction in liver stiffness assessed by magnetic resonance elastography (MRE) | Weeks 0 - 48
  Number of subjects
Proportion of subjects with at least 15% reduction in liver stiffness assessed by magnetic resonance elastography (MRE) | Weeks 0 - 72
  Number of subjects
Change in visceral adipose tissue (L) assessed by magnetic resonance imaging (MRI) | Up to day -20, week 24
  Measured in L
Change in visceral adipose tissue (L) assessed by magnetic resonance imaging (MRI) | Up to day -20, week 48
  Measured in L
Change in visceral adipose tissue (L) assessed by magnetic resonance imaging (MRI) | Up to day -20, week 72
  Measured in L
Change in abdominal subcutaneous adipose tissue (L) assessed by magnetic resonance imaging (MRI) | Up to day -20, week 24
  Measured in L
Change in abdominal subcutaneous adipose tissue (L) assessed by magnetic resonance imaging (MRI) | Up to day -20, week 48
  Measured in L
Change in abdominal subcutaneous adipose tissue (L) assessed by magnetic resonance imaging (MRI) | Up to day -20, week 72
  Measured in L
Change in Body weight (% and kg) | Week 0, week 48
  Measured in kg and %
Change in Body weight (% and kg) | Week 0, week 72
  Measured in kg and %
Change in Waist circumference | Week 0, week 48
  Measured in cm
Change in Waist circumference | Week 0, week 72
  Measured in cm
Change in Body mass index (BMI) | Week 0, week 48
  Measured in kg/sqm
Change in Body mass index (BMI) | Week 0, week 72
  Measured in kg/sqm
Number of treatment-emergent adverse events (TEAEs) | Weeks 0 - 48
  Count of adverse events
Number of treatment-emergent adverse events (TEAEs) | Weeks 0 - 79
  Count and % of adverse events
Number of treatment-emergent hypoglycaemic episodes | Weeks 0 - 48
  Count of episodes
Number of treatment-emergent hypoglycaemic episodes | Weeks 0 - 79
  Count of episodes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (2):
- Germany (2):
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Neuss

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/website/content/how-to-access-clinical-trial-datasets.aspx

REFERENCES:
- [Result] Flint A, Andersen G, Hockings P, Johansson L, Morsing A, Sundby Palle M, Vogl T, Loomba R, Plum-Morschel L. Randomised clinical trial: semaglutide versus placebo reduced liver steatosis but not liver stiffness in subjects with non-alcoholic fatty liver disease assessed by magnetic resonance imaging. Aliment Pharmacol Ther. 2021 Nov;54(9):1150-1161. doi: 10.1111/apt.16608. Epub 2021 Sep 27. PMID 34570916
- [Derived] Andersen G, Plum-Morschel L, Hockings PD, Morsing A, Palle MS, Svolgaard O, Flint A. Clinical Characteristics of a Non-Alcoholic Fatty Liver Disease Population Across the Fibrosis Spectrum Measured by Magnetic Resonance Elastography: Analysis of Screening Data. Adv Ther. 2020 Dec;37(12):4866-4876. doi: 10.1007/s12325-020-01503-x. Epub 2020 Oct 1. PMID 33006125